CLINICAL TRIAL: NCT06344845
Title: Clinical Study of [18F] PM-PBB3 PET Imaging of Tau Protein in Neurodegenerative Diseases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCH-NM-PBB3
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Neurodegenerative Diseases
MeSH Terms: conditions — Neurodegenerative Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: 18F-PBB3 PET/CT (Experimental): Inject18F-PBB3 and then perform PET/CT scan.
  Interventions: Diagnostic Test: 18F-PBB3 PET/CT scan

INTERVENTIONS:
Diagnostic Test: 18F-PBB3 PET/CT scan — Patients with suspected neurodegeneration underwent PET/CT scan after injection of 370MBq (10 mCi)18F-FDG to observe for TAU deposition.

SUMMARY:
In terms of the diagnostic technology of brain neurodegenerative diseases, the injection of positron tracers into the human body, so that it can combine with the corresponding protein, and show its distribution through PET imaging is a mature technology in the industry. At present, several research groups around the world are working on the development and clinical efficacy evaluation of their respective tau imaging agent compounds.This clinical research project intends to display the abnormal changes of tau protein in living brain through [18F]PM-PBB3 PET imaging, which is a second-generation tracer further optimized on the basis of [11C]PBB3, and has the advantages of closer binding to tau protein entanglement and less non-specific binding than similar imaging agents. Better image quality and a wider range of clinical applications.

ELIGIBILITY:
Inclusion Criteria:

* Between 45 and 90 years old; No gender limitation. Brain MRI supported the diagnosis of neurodegeneration, and there was no evidence of other neurological diseases.

Informed consent signed in person by the subject or his legal guardian or caregiver.

Exclusion Criteria:

* Have other serious neurological disorders, or gastrointestinal, cardiovascular, liver, kidney, blood system, tumor, endocrine, respiratory, immune deficiency, and other serious diseases.

Received an experimental drug or device within 1 month (whose efficacy or safety is unclear).

patients who were unwilling to undergo PET/CT scans. pregnancy.

Ages: 49 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Performance | Through study completion, an average of 1 year
  Diagnostic performance including sensitivity, specificity, accuracy

SECONDARY OUTCOMES:
Clinical Stage | Through study completion, an average of 1 year
  Clinical stage changed by 18F-PBB3 PET/CT compared to 18F-FDG PET/CT.

CONTACTS AND LOCATIONS:
Overall Officials: Ruixue Cui, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China